CLINICAL TRIAL: NCT03651804
Title: Radiofrequency Ablation of the Medial Branch Nerve as a Novel Treatment for Posterior Element Pain From Vertebral Compression Fractures
Brief Title: Radiofrequency Ablation: Treatment for Posterior Element Pain From Vertebral Compression Fractures
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting members
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1198963
Record Dates: First submitted 2018-08-14; First posted 2018-08-29 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Vertebral Compression Fracture; Facet Joint Pain
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal; Diphosphonates; Acetaminophen; Physical Therapy Modalities; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): The control group will receive usual care for treatment of vertebral compression fractures, which will consist of but not limited to: physical therapy, opioids, NSAIDs, acetaminophen and bisphosphonates as indicated. They will have the option of crossing over (see "Crossover Group") at twelve weeks.
  Interventions: Drug: Non-steroidal anti-inflammatory drugs; Drug: Bisphosphonates; Drug: Acetaminophen; Behavioral: Physical therapy; Drug: Opioids
- Treatment Group (Active Comparator): The treatment group will receive usual care for treatment and the treatment procedure comprised of the Medial Branch Block and Radiofrequency Ablation. In cases where a medial branch nerve block has confirmed there is pain relief, a radiofrequency ablation is considered. These patients will continue their usual care therapy as well.
  Interventions: Procedure: Radiofrequency ablation of the medial branch nerves; Drug: Non-steroidal anti-inflammatory drugs; Drug: Bisphosphonates; Drug: Acetaminophen; Behavioral: Physical therapy; Drug: Opioids
- Crossover Group (Active Comparator): This group will comprise of patients within the control group who after 12 weeks of usual therapy will have the option of crossing over to the treatment group. Once crossed over, their treatment and course and measurements will be identical to that of the treatment group.
  Interventions: Procedure: Radiofrequency ablation of the medial branch nerves; Drug: Non-steroidal anti-inflammatory drugs; Drug: Bisphosphonates; Drug: Acetaminophen; Behavioral: Physical therapy; Drug: Opioids

INTERVENTIONS:
Procedure: Radiofrequency ablation of the medial branch nerves — A radiofrequency ablation (RFA) is a procedure in which a heat lesion via a needle is created on the nerve that transmits the pain signal in order to interrupt the brain to interrupt the painful signal to the brain. We will target the medial branch nerves.
  Other Names: RFA-MBB
  Arms: Crossover Group; Treatment Group
Drug: Non-steroidal anti-inflammatory drugs — Some of the most commonly used pain medicines in adults. NSAIDs block proteins, called enzymes, in the body that play a role in pain and inflammation. They include aspirin, ibuprofen (Advil, Motrin), naproxen (Aleve), and many other generic and brand name drugs.
  Other Names: NSAID
Drug: Bisphosphonates — A class of drugs that prevent the loss of bone density and are used to treat osteoporosis and similar diseases.
Drug: Acetaminophen — A medicine used to treat pain and fever. It is typically used for mild to moderate pain relief. Commonly known as Tylenol.
  Other Names: Tylenol
Behavioral: Physical therapy — Physical Therapy.
Drug: Opioids — Opioids are narcotics that act on opioid receptors to produce morphine-like effects and medically they are primarily used for pain relief.

SUMMARY:
The purpose of this study is to test the efficacy of radiofrequency ablation of the medial branch nerves (RFA-MBN) in relieving pain and improving physical function in patients with subacute and chronic vertebral compression fractures (VCF).

DETAILED DESCRIPTION:
The study examines a novel approach to treat pain associated with VCFs. The usual care therapy currently involves utilizing physical therapy, non-steroidal anti-inflammatory medications, opioids, and bone re-building medications known as bisphosphonates. A usual treatment plan may include some, if not all the above. There is growing evidence that the posterior spinal elements contribute to pain that patients with VCFs experience. RFA-MBN, which targets these posterior spinal elements, may provide more sustained pain relief and improved physical function compared to usual care for these fractures. The procedure essentially "ablates with heat" the medial branch nerves which send pain signals from the posterior elements to the brain.

Patients will be randomly selected into one of two groups. The treatment group will receive the RFA-MBN procedure along with usual care therapy. The control group will undergo usual care. The control group will have the option to cross over to receive RFA-MBN at a defined interval during the study. There will be follow up visits at various intervals to compare pain relief and function based on various surveys of the treatment, control, and cross-over groups.

ELIGIBILITY:
I• Inclusion

* 18-90 years old
* Male or female
* Age of fracture greater than or equal to 6 weeks
* Single Level Vertebral Compression Fracture
* Vertebral compression fracture Thoraic-9 to Lumbar-5
* NRS >6/10

  • Exclusion
* <18 or >90 yo
* Uncorrectable Coagulopathy
* Multiple Level Vertebral Compression Fractures
* Surgery within 60 days of presentation
* Active infection
* Rhuematologic disease
* Significant neurologic deficit
* Radicular pain
* Chronic low back pain in last year
* Inability to give consent
* Cognitive impairment
* Patients with Ongoing Litigation or Worker's Compensation Cases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) of subjective pain at dedicated Time Frames listed below. | 0 weeks, 1 week, 12 weeks, 6 months
  VAS pain scale (0-10 scale): Overall, at rest, and in bed at night
  The VAS Pain scale is a measure of pain intensity. For pain intensity, the scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).
  Subjects will report their pain prior to the procedure and at dedicated intervals after to assess change in pain intensity they experience.

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire at dedicated time frames listed below to assess change. | 0 weeks, 1 week, 12 weeks, 6 months
  The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The RMQ has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain. It is a series of 24 questions in which a "Yes" response appoints one point. A total score of is 24 possible. Clinical improvement over time can be graded based on the analysis of serial questionnaire scores. If, for example, at the beginningof treatment, a patient's score was 12 and, at the conclusion of treatment, her score was 2 (10 points of improvement), we would calculate an 83% (10/12 x 100) improvement.
QUALEFFO-41 (Quality of Life questionnaire) Scale at dedicated time frames listed below to assess change. | 0 weeks, 1 week, 12 weeks, 6 months
  The Qualeffo-41 is a specific quality of life instrument, which is developed for patients with vertebral compression fractures. This questionnaire comprised of 41 questions, covers main aspects of quality of life: pain, physical functions, social functions, general health and mental health. All answers are standardized so that 1 represents the best and 5 (or 3, or 4) represents the worst quality of life (reverse scores on questions 33, 34, 35, 37, 39, 40). The total score is calculated by summing all answers of questions 1-41. The raw total score ranges from 41 to 205 (or less when some answers are missing) and this is transformed to scores from 0 to 100. The higher the score the poorer the quality of life.
Patient Health Questionnaire (PHQ-9) at dedicated Time Frames listed below. | 0 weeks, 1 week, 12 weeks, 6 months
  The PHQ-9 is a multipurpose instrument for monitoring and measuring the severity of depression. The PHQ-9 incorporates leading major depressive symptoms into a brief self-report tool. It is comprised of a series of 9 questions that assess a series of feelings/symptoms related to clinical depression over the past two weeks and are graded on a scale of 0-3 (gradation of not at all 0 to every day 3). The scores are tallied up for a total score of 0 to 27. The higher the score the greater the severity of the depression.

CONTACTS AND LOCATIONS:
Overall Officials: David Copenhaver, MD, Principal Investigator — UC Davis Medical Center, Department of Anesthesiology and Pain Medicine
Locations (1):
- UC Davis Medical Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boonen S, Van Meirhaeghe J, Bastian L, Cummings SR, Ranstam J, Tillman JB, Eastell R, Talmadge K, Wardlaw D. Balloon kyphoplasty for the treatment of acute vertebral compression fractures: 2-year results from a randomized trial. J Bone Miner Res. 2011 Jul;26(7):1627-37. doi: 10.1002/jbmr.364. PMID 21337428
- [Background] Wardlaw D, Cummings SR, Van Meirhaeghe J, Bastian L, Tillman JB, Ranstam J, Eastell R, Shabe P, Talmadge K, Boonen S. Efficacy and safety of balloon kyphoplasty compared with non-surgical care for vertebral compression fracture (FREE): a randomised controlled trial. Lancet. 2009 Mar 21;373(9668):1016-24. doi: 10.1016/S0140-6736(09)60010-6. Epub 2009 Feb 24. PMID 19246088
- [Background] Klazen CA, Lohle PN, de Vries J, Jansen FH, Tielbeek AV, Blonk MC, Venmans A, van Rooij WJ, Schoemaker MC, Juttmann JR, Lo TH, Verhaar HJ, van der Graaf Y, van Everdingen KJ, Muller AF, Elgersma OE, Halkema DR, Fransen H, Janssens X, Buskens E, Mali WP. Vertebroplasty versus conservative treatment in acute osteoporotic vertebral compression fractures (Vertos II): an open-label randomised trial. Lancet. 2010 Sep 25;376(9746):1085-92. doi: 10.1016/S0140-6736(10)60954-3. Epub 2010 Aug 9. PMID 20701962
- [Background] Buchbinder R, Osborne RH, Ebeling PR, Wark JD, Mitchell P, Wriedt C, Graves S, Staples MP, Murphy B. A randomized trial of vertebroplasty for painful osteoporotic vertebral fractures. N Engl J Med. 2009 Aug 6;361(6):557-68. doi: 10.1056/NEJMoa0900429. PMID 19657121
- [Background] Kallmes DF, Comstock BA, Heagerty PJ, Turner JA, Wilson DJ, Diamond TH, Edwards R, Gray LA, Stout L, Owen S, Hollingworth W, Ghdoke B, Annesley-Williams DJ, Ralston SH, Jarvik JG. A randomized trial of vertebroplasty for osteoporotic spinal fractures. N Engl J Med. 2009 Aug 6;361(6):569-79. doi: 10.1056/NEJMoa0900563. PMID 19657122
- [Background] Johnell O, Kanis JA. An estimate of the worldwide prevalence and disability associated with osteoporotic fractures. Osteoporos Int. 2006 Dec;17(12):1726-33. doi: 10.1007/s00198-006-0172-4. Epub 2006 Sep 16. PMID 16983459
- [Background] Solberg J, Copenhaver D, Fishman SM. Medial branch nerve block and ablation as a novel approach to pain related to vertebral compression fracture. Curr Opin Anaesthesiol. 2016 Oct;29(5):596-9. doi: 10.1097/ACO.0000000000000375. PMID 27548307
- [Background] Bogduk N, MacVicar J, Borowczyk J. The pain of vertebral compression fractures can arise in the posterior elements. Pain Med. 2010 Nov;11(11):1666-73. doi: 10.1111/j.1526-4637.2010.00963.x. PMID 21044256
- [Background] Kim TK, Kim KH, Kim CH, Shin SW, Kwon JY, Kim HK, Baik SW. Percutaneous vertebroplasty and facet joint block. J Korean Med Sci. 2005 Dec;20(6):1023-8. doi: 10.3346/jkms.2005.20.6.1023. PMID 16361816
- [Background] Park KD, Jee H, Nam HS, Cho SK, Kim HS, Park Y, Lim OK. Effect of medial branch block in chronic facet joint pain for osteoporotic compression fracture: one year retrospective study. Ann Rehabil Med. 2013 Apr;37(2):191-201. doi: 10.5535/arm.2013.37.2.191. Epub 2013 Apr 30. PMID 23705113
- [Background] Im TS, Lee JW, Lee E, Kang Y, Ahn JM, Kang HS. Effects of Facet Joint Injection Reducing the Need for Percutaneous Vertebroplasty in Vertebral Compression Fractures. Cardiovasc Intervent Radiol. 2016 May;39(5):740-745. doi: 10.1007/s00270-015-1286-x. Epub 2015 Dec 29. PMID 26714695
- [Background] Mitra R, Do H, Alamin T, Cheng I. Facet pain in thoracic compression fractures. Pain Med. 2010 Nov;11(11):1674-7. doi: 10.1111/j.1526-4637.2010.00953.x. Epub 2010 Oct 1. PMID 21029349
- [Background] Wang B, Guo H, Yuan L, Huang D, Zhang H, Hao D. A prospective randomized controlled study comparing the pain relief in patients with osteoporotic vertebral compression fractures with the use of vertebroplasty or facet blocking. Eur Spine J. 2016 Nov;25(11):3486-3494. doi: 10.1007/s00586-016-4425-4. Epub 2016 Feb 5. PMID 26850264
- [Background] Lord SM, Barnsley L, Wallis BJ, McDonald GJ, Bogduk N. Percutaneous radio-frequency neurotomy for chronic cervical zygapophyseal-joint pain. N Engl J Med. 1996 Dec 5;335(23):1721-6. doi: 10.1056/NEJM199612053352302. PMID 8929263
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- See also: Learn more or sign up for the study here! — https://studypages.com/s/radiofrequency-ablation-heat-therapy-to-reduce-nerve-pain-for-vertebral-compression-fracture-pain-402785/